CLINICAL TRIAL: NCT03835663
Title: Identification of Bacteria Responsible for the the Development of Oesophago-gastric Cancer
Brief Title: The Bacterial Composition of the Stomach in Reflux Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: R18055
Record Dates: First submitted 2019-01-31; First posted 2019-02-08 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: GORD; Oesophageal Cancer; Oesophageal Reflux; Gastric Cancer; Gastro Esophageal Reflux; Oesophageal Carcinoma; Barrett Esophagus; Esophagitis
MeSH Terms: conditions — Esophageal Neoplasms; Gastroesophageal Reflux; Stomach Neoplasms; Barrett Esophagus; Esophagitis | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endoscopic biopsy from gastric mucosa Saliva Liquid gastric content
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with non erosive reflux: Patients with symptoms of reflux but no evidence of oesophagitis or Barretts oesophagus on endoscopy.
  Interventions: Diagnostic Test: No intervention but patients are undergoing an upper GI endoscopy and biopsies for clinical purposes
- Patients with erosive reflux: Patients with symptoms of reflux with evidence of oesophagitis or Barretts oesophagus on endoscopy.
  Interventions: Diagnostic Test: No intervention but patients are undergoing an upper GI endoscopy and biopsies for clinical purposes
- Patients with no reflux: Patients with healthy oesophago-gastric mucosa and no symptoms of reflux.
  Interventions: Diagnostic Test: No intervention but patients are undergoing an upper GI endoscopy and biopsies for clinical purposes

INTERVENTIONS:
Diagnostic Test: No intervention but patients are undergoing an upper GI endoscopy and biopsies for clinical purposes — Standard upper GI endoscopy with biopsies

SUMMARY:
Gastric and oesophageal (OG) cancer associated with poor long term outcome as overall less than 25% of patients survive for more than 5 years due to late recognition of the disease. Growing evidence suggests an important role for bacteria in OG cancer and gastro esophageal reflux disease (GORD) development. About 1 in 10 people suffer from GORD and this one of the most common conditions leading to gastric and oesophageal cancer.

In GORD surgical therapy is the most successful preventing cancer but around 85% of patient experience complications afterwards. Acid suppressing medications are reducing the risk of oesophageal cancer but equally increasing the risk of gastric cancer. They also shorten patients' life expectancy and often fail to provide relief. Analysis of stool samples of patients with GORD demonstrated different gut bacterial compositions to normal and rather resembled the one found in cancer.

There is a clear need to improve the outcome of OG cancer. This could be achieved by identifying bacteria responsible for cancer development in gastric tissue, gastric content and saliva and potentially eliminate them hence avoid the development of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients who deemed necessary for an upper gastro intestinal endoscopy for clinical reasons and consent for additional gastric mucosal biopsies for study purposes

Exclusion Criteria:

* Patients who have upper GI malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with erosive, non-erosive reflux and patients with no symptoms of reflux and healthy upper GI mucosa.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in the bacterial composition of the gastric mucosa between the three groups | Samples are collected on the day of endoscopy following min 6 hours starvation and preserved on -80C
  Bacterias found in the stomach will be identified with 16s RNA analysis. The type of bacterias identified will be compared between the three groups.
Difference in the amount of bacteria of the gastric mucosa between the three previously described groups. | Samples are collected on the day of endoscopy following min 6 hours starvation and preserved on -80C
  Bacterias found in the gastric mucosa will be quantified and compared within the three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare, St Mary's Hospital, Paddington, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No